CLINICAL TRIAL: NCT05394727
Title: Application of Needle-free Injection of Insulin in Pregnant Women With Gestational Diabetes Mellitus
Brief Title: Application of Needle-free Injection of Insulin in Patients With Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NFEC-2019-257
Record Dates: First submitted 2022-05-17; First posted 2022-05-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Injection; Blood Glucose, High; Glycemic Control; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Test group: use needle-free syringe for insulin injection and replace it with conventional insulin pen injection after 2 weeks.
  Control group: use traditional insulin pen injection and replace it with needle-free syringe after 2 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-free injection first group (Experimental): Use needle-free syringe for insulin injection in patients for 2 weeks, then replace it with conventional insulin pen injection for another 2 weeks.
  Interventions: Device: Needle-free injection device, Then traditional insulin pen
- Traditional insulin pen first group (Other): Use conventional insulin pen for insulin injection in patients for 2 weeks, then replace it with needle-free syringe injection for another 2 weeks.
  Interventions: Device: Traditional insulin pen , Then Needle-free injection device

INTERVENTIONS:
Device: Needle-free injection device, Then traditional insulin pen — Patients first received needle-free syringe for insulin injection 3~4 times per day for 2 weeks. After the period of 2 weeks, they then received conventional insulin pen for insulin injection 3~4 times per day for 2 weeks.
  Arms: Needle-free injection first group
Device: Traditional insulin pen , Then Needle-free injection device — Patients first received conventional insulin pen for insulin injection 3~4 times per day for 2 weeks. After the period of 2 weeks, they then received needle-free syringe for insulin injection 3~4 times per day for 2 weeks.
  Arms: Traditional insulin pen first group

SUMMARY:
This study is about the application of needle-free injection device in GDM patients in order to observe the variation of blood glucose and patients' experience compared to the traditional insulin pen injection. To provide evidence for the application of needle-free syringe injection in GDM patients.

DETAILED DESCRIPTION:
This study is a prospective, randomized, unblinded,crossover and controlled clinical trail. The first patient was enrolled on November 1, 2019. The follow-up visit of all enrolled patients in our center will be finished on June 30, 2021. There are two arms in our study : Test Group(IG,n=20) and Control Group(CG,n=20), 40 patients totally.

Test group: "Needle-free injection device, Then traditional insulin pen" Patients first received needle-free syringe for insulin injection 3~4 times per day for 2 weeks. After the period of 2 weeks, they then received conventional insulin pen for insulin injection 3~4 times per day for 2 weeks.

Control group: "Traditional insulin pen , Then Needle-free injection device" Patients first received conventional insulin pen for insulin injection 3~4 times per day for 2 weeks. After the period of 2 weeks, they then received needle-free syringe for insulin injection 3~4 times per day for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients'diagnostic criteria of gestational diabetes mellitus(GDM) is according to the Guidelines for the prevention and control of type 2 diabetes in China (2017 Edition).
* fasting glucose or 2h post prandial glucose was abnormal after 3days' dietary control (fasting glucose ≥ 6.1 mmol/L, or 2h post prandial glucose ≥7.8 mmol/L).
* Aged≥20 years, Han, singleton pregnancy.
* Patients who gave informed consent voluntarily participated in the study, and had regular perinatal examination at our hospital and intended to deliver at our hospital.

Exclusion Criteria:

* Patients with multiple pregnancy or undergoing assisted reproductive technology.
* Patients with polycystic ovary syndrome in preconception.
* Patients with other endocrine metabolic disorders such as gestational hypertension and hyperthyroidism.
* Patients with severe anemia and hypoproteinemia, abnormal liver and kidney function, severe heart failure, respiratory failure and other systemic diseases.
* Patients on long-term medications that affect glucose metabolism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Blood Glucose Indicators to week 4 | Baseline, week 2, week 4
  The blood glucose indicators include fasting blood glucose and blood glucose of 0.5,1,2,3 hours post-meals. Change=(Week 4 blood glucose indicators - Week 2 blood glucose indicators - Baseline blood glucose indicators).
Change from baseline in Plasma insulin concentrations to week 4 | Baseline, week 2, week 4
  The Plasma insulin concentrations include fasting plasma insulin concentration and plasma insulin concentrations of 0.5,1,2,3 hours post-meals. Change=(Week 4 plasma insulin concentrations - Week 2 plasma insulin concentrations - Baseline plasma insulin concentrations).

CONTACTS AND LOCATIONS:
Overall Officials: yaoming Xue, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No